CLINICAL TRIAL: NCT05783661
Title: Randomized Controlled Trial Comparing Conventional Antibiotic Strategies Versus Regimens Guided by Epidemiological Surveillance in Infected Patients With Cirrhosis
Brief Title: Trial Comparing Conventional Antibiotic Strategies Versus Regimens Guided by Epidemiological Surveillance in Infected Patients With Cirrhosis (SURVIC_STUDY)
Acronym: SURVIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eva Bonfill (Other)
Responsible Party: Sponsor-Investigator, Eva Bonfill, Project Manager, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-001858-33
Record Dates: First submitted 2023-02-15; First posted 2023-03-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Decompensated Cirrhosis; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Patients will recieve:
  1. Antibiotic regimens guided by colonization/epidemiological surveillance.
  2. Conventional antibiotic regimens.
Masking Description: The study treatment is not blinded, however the rectal and nasal swabs of the control group will be blinded to the investigator and the participant.
  In all participants, microbiology department will immediately process the samples (swabs) in order to identify a potential colonization by MDR bacteria. Results will be available in the SAP system in patients randomized to the surveillance group but will remained blinded for the clinical investigators in the control group. Blinding will be broken when the patient completes the follow-up period (28 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional antibiotic strategies (Active Comparator): The control group will receive treatment according to the local guidelines of the Hospital Clinic de Barcelona.
  Interventions: Other: Conventional antibiotic strategies
- Regimens guided by epidemiological surveillance (Experimental): The experimental group will receive treatment to the local guidelines of the Hospital Clinic de Barcelona guided by colonization/epidemiological surveillance.
  Interventions: Other: Regimens guided by epidemiological surveillance

INTERVENTIONS:
Other: Conventional antibiotic strategies — Treatment according to the local guidelines of the Hospital Clinic de Barcelona.
  Arms: Conventional antibiotic strategies
Other: Regimens guided by epidemiological surveillance — Treatment according to the local guidelines of the Hospital Clinic de Barcelona guided by colonization/epidemiological surveillance.
  Arms: Regimens guided by epidemiological surveillance

SUMMARY:
Study to comparing conventrional antibiotic strategies versus regimens guided by epidemiological surveillance in infected patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic patients with acute decompensation aged ≥18 years.
2. Proven or suspected bacterial infection requiring antibiotic therapy (diagnosis will be established according to local guidelines, Appendix 1).
3. Signed informed consent or consent given by their legal representatives or close relatives.

Exclusion Criteria:

1. Bacterial infection lasting for > 48 hours.
2. Infection in a critically ill cirrhotic patient (ICU admission). In this population, epidemiological surveillance is standard clinical practice.
3. Evidence of current locally advanced or metastatic malignancy (patients with hepatocellular carcinoma within the Milan criteria and non-melanocytic skin cancer can be included).
4. Pregnant and/or breast-feeding woman.
5. Patients who cannot provide prior informed consent and when there is documented evidence that the patient has no legal surrogate decision-maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Probability/rate of participants of developing antibiotic resistance in both treatment arms at 28 days. | 28 days
  Measured by the appearance of new colonizations and/or infections by MDROs.

SECONDARY OUTCOMES:
Probability of antibiotic resistance development during hospitalization in both treatment arms. | During hospitalization (until discharge), assessed up to day 28.
  Measured by the appearance of new colonizations and/or infections by MDROs.
Rate of antibiotic resistance development during hospitalization in both treatment arms. | During hospitalization (until discharge), assessed up to day 28.
  Measured by the appearance of new colonizations and/or infections by MDROs.
Rate of MDRO colonization during hospitalization and at 28 days in both treatment arms. | During hospitalization (until discharge), assessed up to day 28 and at 28 days.
  Measured by the appearance of new colonications by MDROs.
Probability of MDRO colonization during hospitalization and at 28 days in both treatment arms. | During hospitalization (until discharge), assessed up to day 28 and at 28 days.
  Measured by the appearance of new colonications by MDROs.
Rate of MDRO infection during hospitalization and at 28 days in both treatment arms. | During hospitalization (until discharge), assessed up to day 28 and at 28 days.
  Measured by the appearance of new infections by MDROs.
Probability of MDRO infection during hospitalization and at 28 days in both treatment arms. | During hospitalization (until discharge), assessed up to day 28 and at 28 days.
  Measured by the appearance of new infections by MDROs.
Infection resolution rate with initial and final strategies in both treatment arms. | Through study completion, an average of 28 days
  Measured by the number of infections resolution with initial strategies or final strategies.
Evolution of score ACLF (Acute-on-Chronic Liver Failure) in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of ACLF score. Minimum ACLF score: 6 points. Maximum ACLF score: 18 points. Higher scores means a worse result.
Evolution of score MELD (Model For End-Stage Liver Disease) in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of MELD score. Minimum MELD score: 6 points. Maximum MELD score: 40 points. Higher scores means a worse result.
Evolution of score Child-Pugh in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of Child -Pugh score. Minimum Child-Pugh score: 5 points. Maximum Child-Pugh score: 15 points. Higher scores means a worse result.
Evolution of score CLIF-OF (Liver Failure Consortium - Organ Failure) in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of CLIF-OF score. Minimum CLIF-OF score: 6 points. Maximum CLIF-OF score: 18 points. Higher scores means a worse result.
Evolution of score CLIF-C AD (Chronic Liver Failure Consortium - non-ACLF patients with Acute Decompensation) in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of CLIF-C AD score.
  Minimum CLIF-C AD score: 6 points. Maximum CLIF-C AD score: 18 points. Higher scores means a worse result.
Evolution of score CLIF-C ACLF (Chronic Liver Failure Consortium - Acute-on-Chronic Liver Failure) in both treatment arms. | Through study completion, an average of 28 days
  Measured by the result of CLIF-C ACLF score. Minimum CLIF-C ACLF score: 6 points. Maximum CLIF-C ACLF score: 18 points. Higher scores means a worse result.
Days of admission to the ICU if needed. | Through study completion, an average of 28 days
  Measured by the days of admission to the ICU.
Days of life support (dialysis, vasopressors, and mechanical ventilation) if needed. | Through study completion, an average of 28 days
  Measured by the days of life support.
Days of hospital stay | Through study completion, an average of 28 days
  Measured by the days of hospital stay.
Number of rehospitalizations. | Through study completion, an average of 28 days
  Measured by the number of rehospitalizations.
Antibiotics consumption | Through study completion, an average of 28 days
  Measured by the days of antibiotics consumption.
Antibiotics consumption | Through study completion, an average of 28 days.
  Measured by dose of antibiotics.
Antibiotics consumption | Through study completion, an average of 28 days
  Measured by type of antibiotics.
Health costs | Through study completion, an average of 28 days
  Measured by the cost of antibiotic, cost of hospital/ICU stay and of organ support(s).
Proportion of participants with antibiotic-related AE, SAEs, SUSARs and other SAEs. | Through study completion, an average of 28 days
  Measured by the number of participants with antibiotic-related AE, SAEs, SUSARs and other SAEs.
Hospital survival | During hospitalization (until discharge), assessed up to day 28.
  Number of survival participants
28-day survival | 28 days
  Number of survival participants

CONTACTS AND LOCATIONS:
Locations (1):
- Eva Bonfill, Barcelona, Spain